CLINICAL TRIAL: NCT07063550
Title: Identification of Paraneoplastic and Intratumoral Microplastics in Colorectal Cancer and Their Association Analysis With Macrogenomics and Metabolomics
Brief Title: Microplastics in Paraneoplastic and Intratumoral for Colorectal Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Dong Peng (Other)
Responsible Party: Sponsor-Investigator, Dong Peng, Principal Investigator, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: 2024-531-01
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer (MSI-H); Microplastic Exposure
Keywords: colorectal cancer; microplastic; Paraneoplastic; Genomics; Metabolomics
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- the colorectal cancer group: patients diagnosed with colorectal cancer
  Interventions: Other: exposure to microplastic

INTERVENTIONS:
Other: exposure to microplastic — Microplastic content in cancerous and paracancerous tissues

SUMMARY:
The objective of this study is to identify and characterize microplastics present in peritumoral and intratumoral tissues of colorectal cancer patients, and to investigate their associations with gut microbiome composition and metabolic profiles. By integrating microplastic analysis with metagenomic and metabolomic data, we aim to explore the potential impact of environmental microplastic exposure on tumor microenvironment alterations, microbial dysbiosis, and metabolic reprogramming in colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old) with histologically confirmed colorectal adenocarcinoma.
* Undergoing elective radical colorectal cancer resection at the study hospital.
* No prior chemotherapy, radiotherapy, or targeted therapy before surgery.
* Availability of both tumor tissue and adjacent normal (peritumoral) tissue samples during surgery.
* Willingness to provide stool and/or blood samples for metagenomic and metabolomic analysis.
* Ability to understand the study procedures and provide written informed consent.

Exclusion Criteria:

* Patients with a history of other malignancies within the past 5 years.
* Emergency surgery due to obstruction, perforation, or bleeding.
* Inadequate sample quality or volume for microplastic, metagenomic, or metabolomic analysis.
* Presence of chronic inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis).
* Use of antibiotics, probiotics, or prebiotics within 4 weeks prior to sample collection.
* Pregnant or breastfeeding women.
* Refusal or inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with colorectal cancer and received rectal cancer surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
genomics | Blood specimens were obtained within one week prior to surgery.
  Genomics was tested by preoperative blood specimens.

SECONDARY OUTCOMES:
metabolomics | Blood specimens were obtained within one week prior to surgery.
  Metabolomics was tested by preoperative blood specimens.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Due to the requirements of the Ethics Committee, it was not permitted to make the acquired data public.